CLINICAL TRIAL: NCT00377273
Title: An Open-Label 18-Month Safety Study of Fluorouracil Cream 0.5% for the Treatment of Actinic Keratoses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DL6025-0201
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

INTERVENTIONS:
Drug: fluorouracil cream 0.5%

SUMMARY:
This study is being undertaken to: 1. assess the safety of fluorouracil cream for the treatment of actinic keratoses ("AKs") on other common skin surface areas (e.g., posterior scalp, ears, neck, lips, arms and hands); 2. collect additional post-treatment safety data on fluorouracil cream applied to the face (including anterior scalp, if applicable); 3. assess the incidence of recurrence of AKs on the face; and 4. assess the need for re-treatment with fluorouracil cream to the face.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

INCLUSION CRITERIA:

* Patients must give written informed consent;
* Patients must have at least 5 visible and/or palpable AKs on the posterior scalp, ears, neck, lips, arms and/or hands (across all other body sites) and an additional 5 visible and/or palpable AKs on the face (including anterior scalp, if applicable);
* Female patients must be post-menopausal for at least one year, or have had a hysterectomy, or have had a tubal ligation, or use oral/systemic contraceptives, an intrauterine device (IUD) or Norplant starting at least 28 days prior to study entry and throughout the study. Female patients of childbearing potential must have a negative urine pregnancy test prior to the first application of test medication
* Patients must be compliant and willing to return to the study site for designated follow-up visits.

EXCLUSION CRITERIA:

* Pregnant or lactating females;
* Patients with a current skin condition on the face, scalp, ears, neck, lips, arms and/or hands that could confound the study, including basal cell and squamous cell carcinomas;
* Patients with a known allergy to any ingredients of the test drug formulations;
* Patients with known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency;
* Patients whose activities involve excessive or prolonged exposure to sunlight;
* Patients who use a tanning parlor;
* Patients treated with other topical agents for the treatment of actinic keratosis in the designated treatment area within 5 months prior to the start of the study are prohibited;
* Patients who have had liquid nitrogen treatment for AKs within 4 weeks prior to study start in the designated treatment area;
* History of drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2003-11; Study Completion 2005-10

PRIMARY OUTCOMES:
The reduction in Actinic Keratosis lesion counts on other body sites from pretreatment to post-treatment and AK clearance of other body site lesions for Treatment Cycle 1.

SECONDARY OUTCOMES:
The reduction in Actinic Keratosis lesion counts of the face (including anterior scalp, if applicable) from pretreatment to post-treatment and AK clearance of facial lesions for each Treatment Cycle
The recurrence of facial lesions at 12 and 18 months post initial treatment, and the need for re-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, MT, ASCP, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States